CLINICAL TRIAL: NCT06552195
Title: Hologram-Based Augmented Reality in Learning Anatomy: The TEACHANATOMY Randomized Cross-over Trial
Brief Title: Augmented Reality in Learning Anatomy: The TEACHANATOMY Randomized Cross-over Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Collaborators: ETH Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: TEACHANATOMY 2.0
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Augmented Reality; Anatomy Education
Keywords: Anatomy teaching; Augmented reality; Magic leap
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: outcomes (knowledge test, adverse health symptoms and user experience) will be assessed blindly
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shoulder anatomy with augmented reality (AR) , hips anatomy with traditional learning (TL) (Experimental): Participants first learn the shoulder anatomy with AR. After a washout period of three weeks, they will learn the hips anatomy with traditional Learning (TL) methods
  Interventions: Other: learning with augmented reality; Other: learning with traditional methods
- Traditional learning (TL) group. (Active Comparator): Participants first learn the shoulder anatomy with Traditional learning methods. After a washout period of three weeks, they will learn the hips anatomy with augmented reality (AR)
  Interventions: Other: learning with augmented reality; Other: learning with traditional methods

INTERVENTIONS:
Other: learning with augmented reality — Study presentation: participants will be given a 10-minute general introduction on the study followed by a 20 minutes tutorial to introduce the HoloLens 2 and the TEACHANATOMY learning platform.
  * Study session: The study session consists of three learning blocks of approximately 20 minutes each, plus a repetition block to assess the acquired knowledge. During the study session participants will be given no time constraints and free breaks.
  * Assessment test: Participants will be assessed with a 30 minutes knowledge assessment test at the end of the study and after three months.
  * Final questionnaire: At the end of the study session participants will be given a questionnaire to assess adverse health symptoms and user experience.
Other: learning with traditional methods — * Study presentation: participants will be given a 10-minute general introduction on the study followed by a presentation to introduce the study session.
  * Study session: The study session consists of the learning resources most used by students: specific sections from four different neuroanatomy books, access to two websites, two 3D videos, and two online learning programs. During the study session participants will be given no time constraints and free breaks.
  * Assessment test: Participants will be assessed with a 30 minutes knowledge assessment test at the end of the study and after three months.
  * Final questionnaire: At the end of the study session participants will be given a questionnaire to assess adverse health symptoms and user experience

SUMMARY:
Cadaver use in anatomy education is undergoing several limitations in many universities, due to high costs, time constraints and supply difficulties. As alternatives to cadaver dissections, new teaching methods based on visual technologies, such as augmented reality (AR), are being implemented worldwide.

Augmented reality (AR), based on virtual interactive 3-dimensional elements (holograms) overlaid in the real-world, represents a promising alternative to explore the human body. In this study, we will test the efficacy of AR as an alternative teaching method in anatomy education by comparing traditional learning methods based on 2-dimensional (2D) images, videos, and online learning programs with the novel AR learning module The primary endpoint will consist of the score in the final theoretical and practical knowledge tests, assessed at two timepoints: immediately after the study session and after 3 months.

Secondary endpoints will include adverse health symptoms and user experience, assessed immediately after the study session.

DETAILED DESCRIPTION:
Cadaver use in anatomy education is undergoing several limitations in many universities, due to high costs, time constraints and supply difficulties. As alternatives to cadaver dissections, new teaching methods based on visual technologies, such as augmented reality (AR), are being implemented worldwide.

Augmented reality (AR), based on virtual interactive 3-dimensional elements (holograms) overlaid in the real-world, represents a promising alternative to explore the human body. In this study, we will test the efficacy of AR as an alternative teaching method in anatomy education. Our hypothesis is that learning with AR is more efficient than traditional learning methods.

Preparation: We will prepare 2 fresh-frozen cadaveric specimens to allow visualization of anatomical structure of the shoulder and hips. The cadavers will be obtained from a human body donated for university teaching activities. Using a digital single-lens reflex camera, we will acquire several images. These images will be then converted into a 3D model by the ROCS team at Balgrist University Hospital and optimized for use with the Magic Leap AR headset.

Procedure: Participants (approx. 300) will be randomly assigned to the AR or the traditional learning (TL) group. Each participant will learn one anatomy module with traditional learning methods, which will include books, access to websites, 3D videos, and online learning programs, and one module with the AR-based learning program. The two modules will be administered approximately 3 weeks apart.

Group A: Shoulder anatomy with traditional learning methods and hips anatomy with AR based 3D program.

Group B: Shoulder anatomy with AR based 3D program and hips anatomy with traditional learning methods.

The primary endpoint will consist of the score in the final theoretical and practical anatomy tests, assessed at two timepoints: immediately after the study session and after 3 months.

Secondary endpoints include adverse health symptoms, assessed with a Likert scale survey, and user experience, evaluated using an adapted NASA Task Load Index scale plus additional questions.

ELIGIBILITY:
Inclusion Criteria:

* Medical students attending the 1st or 2nd year of undergraduate medical education
* Must not have prior anatomical education

Exclusion Criteria:

* Epilepsy
* Binocular vision disorder such as strabismus
* Current head and/or neck injuries
* Inflammation of the scalp and/or eye
* Amputations or partial amputations of the hands

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
knowledge test | immediately after the study session, day 1, and after three months
  The primary outcome will consist of the score in the final theoretical and practical tests. The theoretical test consists of single and multiple-choice questions in which participants will be required to recognize and name the different anatomical structures of the hips or shoulder and their function. In the practical part, participants will be required to mark specific anatomical structures in a 3D-printed anatomical skull model. The duration of the test will be of approximately 30 minutes.

SECONDARY OUTCOMES:
adverse health symptoms | Immediately after the knowledge test, Day 1
  Secondary outcomes will include adverse health symptoms, evaluated with a questionnaire to assess presence and severity of general symptoms (General discomfort, Fatigue, Headache, Dizziness, Nausea, Concentration problems, Disorientation, Neck stiffness/neck pain, No symptoms) and eye-related symptoms (Blurred vision, Difficulty focusing, Double-vision, Dry eyes No symptoms). Presence and severity of symptoms will be rated on a Likert scale from 1 (almost imperceptible) to 10 (extreme).
User experience | Immediately after the Adverse health symptoms, Day 1
  User experience will be assessed using an adapted NASA Task Load Index (5 questions, range, 1-10, with lower scores indicating lower cognitive workload) plus additional 10-point Likert scale and open-ended questions in which participants will be asked to rank their comfort with the material and hardware and the teaching effectiveness of the software or of the traditional learning methods to learn anatomy

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Zingg, MD, Principal Investigator — Balgrust University Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stromberga Z, Phelps C, Smith J, Moro C. Teaching with Disruptive Technology: The Use of Augmented, Virtual, and Mixed Reality (HoloLens) for Disease Education. Adv Exp Med Biol. 2021;1317:147-162. doi: 10.1007/978-3-030-61125-5_8. PMID 33945136
- [Background] Bolek KA, De Jong G, Henssen D. The effectiveness of the use of augmented reality in anatomy education: a systematic review and meta-analysis. Sci Rep. 2021 Jul 27;11(1):15292. doi: 10.1038/s41598-021-94721-4. PMID 34315955
- [Background] Chytas D, Johnson EO, Piagkou M, Mazarakis A, Babis GC, Chronopoulos E, Nikolaou VS, Lazaridis N, Natsis K. The role of augmented reality in Anatomical education: An overview. Ann Anat. 2020 May;229:151463. doi: 10.1016/j.aanat.2020.151463. Epub 2020 Jan 21. PMID 31978568
- [Background] Curran VR, Xu X, Aydin MY, Meruvia-Pastor O. Use of Extended Reality in Medical Education: An Integrative Review. Med Sci Educ. 2022 Dec 19;33(1):275-286. doi: 10.1007/s40670-022-01698-4. eCollection 2023 Feb. PMID 36569366
- [Background] Gsaxner C, Li J, Pepe A, Jin Y, Kleesiek J, Schmalstieg D, Egger J. The HoloLens in medicine: A systematic review and taxonomy. Med Image Anal. 2023 Apr;85:102757. doi: 10.1016/j.media.2023.102757. Epub 2023 Jan 21. PMID 36706637
- [Background] McBain KA, Habib R, Laggis G, Quaiattini A, M Ventura N, Noel GPJC. Scoping review: The use of augmented reality in clinical anatomical education and its assessment tools. Anat Sci Educ. 2022 Jul;15(4):765-796. doi: 10.1002/ase.2155. Epub 2022 Jan 19. PMID 34800073
- [Background] Moro C, Birt J, Stromberga Z, Phelps C, Clark J, Glasziou P, Scott AM. Virtual and Augmented Reality Enhancements to Medical and Science Student Physiology and Anatomy Test Performance: A Systematic Review and Meta-Analysis. Anat Sci Educ. 2021 May;14(3):368-376. doi: 10.1002/ase.2049. Epub 2021 Feb 26. PMID 33378557
- [Background] Navab N, Martin-Gomez A, Seibold M, Sommersperger M, Song T, Winkler A, Yu K, Eck U. Medical Augmented Reality: Definition, Principle Components, Domain Modeling, and Design-Development-Validation Process. J Imaging. 2022 Dec 23;9(1):4. doi: 10.3390/jimaging9010004. PMID 36662102
- [Background] Stojanovska M, Tingle G, Tan L, Ulrey L, Simonson-Shick S, Mlakar J, Eastman H, Gotschall R, Boscia A, Enterline R, Henninger E, Herrmann KA, Simpson SW, Griswold MA, Wish-Baratz S. Mixed Reality Anatomy Using Microsoft HoloLens and Cadaveric Dissection: A Comparative Effectiveness Study. Med Sci Educ. 2019 Nov 15;30(1):173-178. doi: 10.1007/s40670-019-00834-x. eCollection 2020 Mar. PMID 34457656
- [Background] Uruthiralingam U, Rea PM. Augmented and Virtual Reality in Anatomical Education - A Systematic Review. Adv Exp Med Biol. 2020;1235:89-101. doi: 10.1007/978-3-030-37639-0_5. PMID 32488637
- [Result] Moro C, Stromberga Z, Raikos A, Stirling A. The effectiveness of virtual and augmented reality in health sciences and medical anatomy. Anat Sci Educ. 2017 Nov;10(6):549-559. doi: 10.1002/ase.1696. Epub 2017 Apr 17. PMID 28419750
- See also: Magic Leap headsets devise — https://www.magicleap.com/en-gb